CLINICAL TRIAL: NCT05050721
Title: Natural History of Non Alcoholic Fatty Liver Disease and Predictors of Advanced Fibrosis
Status: Withdrawn | Type: Observational
Why Stopped: PI decided to stop the study
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 043.HEP.2019.D
Record Dates: First submitted 2020-09-22; First posted 2021-09-20 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Non-alcoholic Steatohepatitis (NASH)
Keywords: Chronic liver disease, steatosis, inflammation, fibrosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Inflammation; Fibrosis | interventions — Postmortem Imaging; High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: CT imaging — clinical, radiological and biochemical parameters associated with disease progression
  Other Names: ultrasound, fibroscan, MR-Elastrography, liver biopsy

SUMMARY:
The prevalence of non-alcoholic fatty liver disease (NAFLD ) in the American population is approximately 30% in adults and 10% in children, making it the most common. Cause of chronic liver disease in the United States. Although the majority of patients with NAFLD have a benign clinical course, the development of non-alcoholic steatohepatitis (NASH ), with necro-inflammation and progressive fibrosis, increases the risk for development of cirrhosis and its complications. Among patients with NASH, approximately 28% develop cirrhosis over an 8-year follow-up period. NASH and advanced fibrosis is associated with increased morbidity and mortality among those patients with advanced histologic severity such as NASH and fibrosis the gold standard for diagnosing and staging NAFLD is liver biopsy. Liver biopsy is associated with costs and risks that make it impractical for generalized use in a condition that affects such a high portion of the population. Furthermore, liver biopsy is also limited by significant sampling error in NAFLD. Thus, there is a pressing need for accurate non-invasive predictors of NAFLD that would also allow differentiation of those subjects at higher risk of disease progression. At present, in the clinical setting, some demographic factors, blood tests, and imaging studies can be used to predict a higher risk of disease in patients being evaluated for NAFLD. These predictors, however, are of limited sensitivity and specificity compared with liver biopsy. The development and validation of accurate predictors and scoring systems to identify patients at higher risk for NASH and fibrosis would allow identification of subjects who would benefit the most from liver biopsy and potentially help monitor disease

DETAILED DESCRIPTION:
It is a retrospective chart review study. All Methodist Dallas Medical Center (MDMC) patients with fatty liver diseases meeting the inclusion and exclusion criteria as mentioned below will be included in the study. Charts from Jan 2000 - Jan 2019 will be reviewed for data collection.

Data variables: age, weight, Height , BMI, gender, AST, ALT, Bilirubin, albumin, Alkaline phosphatase, WBC, PLT, Hb, sodium, potassium, creatinine, ferritin, insulin, glucose , HDL, LDL,VLDL, cholesterol, triglyceride. CT imaging, ultrasound findings, fibroscan, MR-Elastrography, liver biopsy results, presence of comorbidities like diabetes, hypertension and dyslipidemia

ELIGIBILITY:
Inclusion Criteria:

* All patients both male and female greater than 18 years with radiologic or histologic evidence of fatty liver will be included in the study.

Exclusion Criteria:

* Patients with history of fatty liver less than 18 years of age.
* Patient's with fatty liver consuming alcohol up to greater than one drink per day.
* All fatty liver patients with other chronic liver disease such as hepatitis B, hepatitis C, primary biliary cirrhosis, primary biliary cholangitis, autoimmune hepatitis, alpha one antitrypsin disease or Wilsons disease superimposed on fatty liver disease.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: chronic liver disease registry and EPIC at liver institute and MDMC. All patients meeting the inclusion criteria will be included for the retrospective chart based study from Jan 2000 - Jan 2019.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2021-08-10 (Estimated); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Risk factor (Age) | 1 year
  Age will be measured in years
Risk factor (BMI) | 1 year
  Weight and height will be measured to determine BMI. it will be measured in kg/m^2.

CONTACTS AND LOCATIONS:
Overall Officials: Mangesh Pagadala, M.D., Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- The Liver Institute at Methodist Dallas Medical Center, Irving, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided